CLINICAL TRIAL: NCT04463277
Title: Therapeutic Effects of Time Restricted Feeding and Calorie Restriction in Patients With Prediabetes and Diabetes
Brief Title: A Comparison Between the Effects of Conventional Diets vs Intermittent Fasting Diabetic and Pre-diabetic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Usman Bin Hameed (Other)
Collaborators: World Health Organization (Other)
Responsible Party: Sponsor-Investigator, Usman Bin Hameed, Principal Investigator, Aga Khan University
Organization: Aga Khan University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IFCR-186
Record Dates: First submitted 2020-07-05; First posted 2020-07-09 (Actual); Last update posted 2021-06-08 (Actual); Status verified 2021-06

CONDITIONS: Diabetes Mellitus, Type 2; PreDiabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Prediabetic State | interventions — Caloric Restriction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Calorie Restriction (Experimental)
  Interventions: Behavioral: Calorie Restriction
- Time Restricted Feeding (Experimental)
  Interventions: Behavioral: Time Restricted Feeding
- Time Restricted Feeding with Calorie Restriction (Experimental)
  Interventions: Behavioral: Time Restricted Feeding with Calorie Restriction
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Calorie Restriction — Participants assigned to this arm to consume food at a caloric deficit of 500 calories per day.
  Arms: Calorie Restriction
Behavioral: Time Restricted Feeding — Participants assigned to this arm to consume food at maintenance calories (calories required per day to maintain weight, calculated based on height, weight and physical activity using the MyFitnessPal application) within an 8-hour window during daylight hours.
  Arms: Time Restricted Feeding
Behavioral: Time Restricted Feeding with Calorie Restriction — Participants assigned to this arm to consume food at a caloric deficit of 500 calories per day within an 8-hour window during daylight hours.
  Arms: Time Restricted Feeding with Calorie Restriction

SUMMARY:
This research aims to find an effective dietary intervention among the Pakistani population. According to WHO, diabetes is on the rise in developing countries; the current prevalence among the Pakistani population is 11.2% which is expected to increase in the coming years which is in line with the similar documented trend in neighboring south Asian countries.3,11 Since, ethnic south Asians carry a greater risk for developing T2D at a younger age and along with the complications associated with diabetes due to its chronicity, this poses a significant threat and an increased disease burden on the health care system.11

This will be the first trial conducted on determining the efficacy of caloric restriction in a subset of Pakistani population. There is limited inconsistent data on the efficacy of time-restricted feeding, however, this will help elucidate if it does lead to positive effects on the bio-health markers. One of the major hurdles in caloric restriction is patient compliance, therefore, one of the intervention group will be used to determine if TRF with caloric restriction helps improve the patient's compliance and produces significant results. If such an intervention is effective in inducing weight loss it can also be applied for other overweight patients. Eventually, it will help in countering the rising obesity in the region.

The ultimate purpose of the knowledge obtained is to find a patient friendly, novel and therapeutic dietary intervention which will help in limiting the rise in T2D patients. It'll help in introducing an effective lifestyle intervention to promote health, which will reduce the dependence on pharmacological therapies, as well as, in the long-term reduce burden on the health care system.

The information obtained can provide framework for new guidelines in helping the patients to lose weight, which can be utilized by the government to increase general awareness which will help prevent diseases linked to obesity. In light of the randomized controlled trial, the primary health physicians can educate and increase awareness regarding the different dietary interventions the patients can utilize which will help increase the number of options for the patients. Social media platforms can be utilized due to their extended outreach for the transmission of accurate information to the general population.

ELIGIBILITY:
Inclusion Criteria:

* Glycemic values belonging to diabetes or prediabetes category.
* Weight stable for at least 6 months prior to start of study.
* Ability to understand English and use English language mobile applications.

Exclusion Criteria:

* Pregnant or breastfeeding women.
* Diabetics taking insulin or sulfonylureas.
* Smokers.
* History of cardiovascular disease.
* History of psychiatric or eating disorders.
* History of hypoglycemic episodes.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-05-15 (Actual); Study Completion 2021-05-15 (Actual)

PRIMARY OUTCOMES:
Weight | 12 weeks
  Change in participants' weight.
FBS | 12 weeks
  Change in participants' fasting plasma glucose levels.
HbA1c | 12 weeks
  Change in percentage of glycated hemoglobin HbA1c in the participants' plasma.
OGTT | 12 weeks
  Change in participants' response to an oral glucose load.
Serum Lipid Profile. | 12 weeks
  Change in participant's serum lipid levels, including cholesterol, LDL, HDL and triglycerides.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Nadeem, M.B.B.S, M.D., Principal Investigator — The Aga Khan University Hospital
Locations (1):
- The Aga Khan University Hospital, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No